CLINICAL TRIAL: NCT06402487
Title: Propionic Acid in Multiple Sclerosis - a Placebo-controlled Randomized Double-blinded Clinical Trial
Brief Title: Propionic Acid in Multiple Sclerosis
Acronym: MADAI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Tobias Moser, Principal Investigator, Salzburger Landeskliniken
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1026/2024
Record Dates: First submitted 2024-04-29; First posted 2024-05-07 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Propionic Acid; Progression; Disability; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Disease Progression; Fatigue | interventions — propionic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propionic acid 1000 mg (Active Comparator)
  Interventions: Dietary Supplement: Propionic acid 1000 mg capsule
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Propionic acid 1000 mg capsule — Patients will be assigned to propionic acid or placebo as add on MS treatment.
  Arms: Propionic acid 1000 mg
Dietary Supplement: Placebo — Patients will be assigned to propionic acid or placebo as add on MS treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the superiority of propionic acid over placebo as add on treatment in multiple sclerosis (MS).

DETAILED DESCRIPTION:
This is a single-center, double-blinded, randomized trial. One hundred multiple sclerosis (MS) patients will be randomly assigned in a 2:1 ratio to receive either 100 mg of propionic acid or a placebo over a period of 90 days. Outcome measures will encompass NfL and GFAP levels, fatigue scores, quality of life assessments, and physical examinations. Additionally, subgroup analysis will involve the evaluation of MRI and MEG data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis (MS)
* Clinically and radiologically stable MS in the previous 3 months
* Age between 18 and 60 years
* Positive finding for oligoclonal bands (OCBs)
* Written consent
* Blood collection at the beginning and end of the study for routine parameter examination as well as sample preservation (especially for measuring propionic acid levels)
* Negative pregnancy test for female participants of childbearing age

Exclusion Criteria:

* Existing propionic acid supplementation
* Change in disease-modifying therapy (DMT) in the previous 4 weeks
* Existing severe systemic diseases
* Presence of other concomitant structural nerve diseases (e.g., polyneuropathy, brain tumor, strokes)
* High JCV titer under Natalizumab

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Serum neurofilament light chain (NfL) | 90 days
  assessed as pg/ml
Serum glial fibrillary acid protein (GFAP) | 90 days
  assessed as pg/ml

SECONDARY OUTCOMES:
Fatigue Scale for Motor and Cognitive Functions (FSMC) | 90 days
  Fatigue Score, Questionnaire
Walking test, 10 meters distance | 90 days
  assessed as seconds
cerebral MRI | 90 days
  number of rim lesions; subgroup analysis
36-Item Short Form Health Survey (SF-36) | 90 days
  Quality of Life, Questionnaire
Magnetoencephalography (MEG) | 90 days
  Assessing neuronal slowing proposed as a marker of cognitive impairment in MS; Subgroup analysis
9-hole peg test | 90 days
  assessed in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Salzburger Landeskliniken, Salzburg, Salzburg, Austria

REFERENCES:
- [Background] Duscha A, Gisevius B, Hirschberg S, Yissachar N, Stangl GI, Dawin E, Bader V, Haase S, Kaisler J, David C, Schneider R, Troisi R, Zent D, Hegelmaier T, Dokalis N, Gerstein S, Del Mare-Roumani S, Amidror S, Staszewski O, Poschmann G, Stuhler K, Hirche F, Balogh A, Kempa S, Trager P, Zaiss MM, Holm JB, Massa MG, Nielsen HB, Faissner A, Lukas C, Gatermann SG, Scholz M, Przuntek H, Prinz M, Forslund SK, Winklhofer KF, Muller DN, Linker RA, Gold R, Haghikia A. Propionic Acid Shapes the Multiple Sclerosis Disease Course by an Immunomodulatory Mechanism. Cell. 2020 Mar 19;180(6):1067-1080.e16. doi: 10.1016/j.cell.2020.02.035. Epub 2020 Mar 10. PMID 32160527